CLINICAL TRIAL: NCT03982524
Title: Enriching Cognitive-Behavioral Therapy With Emotion Regulation Training in Patients With Chronic Multiple Somatoform Symptoms (ENCERT): A 3-Year Follow-up of a Randomized Controlled Trial
Brief Title: CBT Enriched With Emotion Regulation Training for Multiple Somatoform Symptoms (ENCERT) - A 3-year Follow-up
Acronym: ENCERT-3YFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENCERT-042017; KL 3132/2-4 (Other Grant/Funding Number: German Research Foundation)
Record Dates: First submitted 2019-06-08; First posted 2019-06-11 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Somatic Symptom Disorder (DSM-5)
Keywords: somatoform symptoms; somatic symptoms; somatoform disorder; somatic symptom disorder; cognitive-behavioral therapy; emotion regulation training; 3-year follow-up
MeSH Terms: conditions — Medically Unexplained Symptoms; Somatoform Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT complemented with emotion regulation training (Experimental): ENCERT contains 1) psychoeducation (session1), 2) relaxation techniques for coping with stress (sessions 2-4), 3) non-judgmental awareness of body perceptions, (sessions 5-7), 4) modifying illness behavior and accepting unpleasant body perceptions (sessions 8-13), 5) attention defocusing on positive perceptions plus emotional self-support (sessions 14- 15), 6) analyzing interpretation processes to understand situational cues (sessions 16-17), and 7) change of behavior and interpretations (sessions 18-20). The innovative elements of ENCERT are: improving the awareness for the association of somatic symptoms with emotions, learning nonjudgmental awareness and acceptance of unpleasant body perceptions, achieving high-frequent skill exercising with the emotion regulation audio training.
  Interventions: Behavioral: Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms
- Cognitive behavior therapy (CBT) (Active Comparator): This arm is based on conventional cognitive-behavioral therapy that can be considered the current "treatment of choice", being the only intervention with an evidence grade 1a (Kroenke, 2007). As such, it presents the reference of efficacy and safety for new regimen. The strictly manualized program includes the following components focusing on the special needs of chronic somatoform patients: psychoeducation providing a framework for psychotherapy, attention defocusing, reduction of over-interpretation of symptoms, increase of physical activity, stress reduction.
  Interventions: Behavioral: Cognitive-behavioral therapy for patients with multiple somatoform symptoms

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms — Cognitive-behavioral therapy + emotion regulation training for patients with multiple somatoform symptoms: 20 weekly sessions individual therapy (à 50 minutes)
  Arms: CBT complemented with emotion regulation training
Behavioral: Cognitive-behavioral therapy for patients with multiple somatoform symptoms — Cognitive-behavioral therapy for patients with multiple somatoform symptoms: 20 weekly sessions individual therapy (à 50 minutes)
  Arms: Cognitive behavior therapy (CBT)

SUMMARY:
The purpose of this study is to evaluate whether 3 years after the end of therapy cognitive-behavioral therapy complemented with strategies from emotion regulation training leads to better improvement in somatic symptoms and comorbid problems in patients with chronic multiple somatoform symptoms than cognitive behavioral therapy alone.

DETAILED DESCRIPTION:
Somatic symptoms not caused by a known biomedical condition ("somatoform disorders") are highly prevalent, involve a high risk of chronicity, are one of the major reasons for doctor visits, and are a tremendous burden for health care systems. Despite the economic relevance, research activities are disproportionately low. The only intervention with an evidence grade I is cognitive behavioral therapy (CBT). However, average effect sizes for CBT in somatization syndromes are only moderate (Cohen's d < 0.5), and more powerful interventions are needed.

There is convincing evidence that patients with somatoform disorders have emotion regulation deficits, which are not addressed by current CBT approaches. We conducted a randomized controlled trial in which we compared a conventional CBT for patients with chronic multiple somatoform symptoms with CBT complemented with emotion regulation techniques (ENCERT; see ClinicalTrials.gov ID: NCT01908855). Previous interventional studies have mainly focused on acute effects and rarely include follow-up periods > 2 years after the end of therapy. The primary goal of the proposed project is to investigate whether effects that were demonstrated for both treatments in our previous randomized controlled trial can be maintained until 3 years after the end of therapy.

This study is based on the intention-to-treat (ITT) sample (N=255 patients) of our previous randomized controlled trial (ClinicalTrials.gov ID: NCT01908855). Patients were primarily recruited via referrals by primary care doctors. After a screening phase baseline assessments with different self- and clinician rating scales (see Outcome Measures) followed. Participants who fulfilled the eligibility criteria were randomized to one of the two study arms: cognitive behavioral therapy vs. cognitive-behavioral therapy complemented with emotion regulation strategies. The post assessment took place after the 20th therapy session and at a follow-up at six months after post treatment. In the current project all randomized patients will be reassessed 3 years after the end of therapy.

Different methods were applied to prevent bias and to assure a high quality level of the current study. Data handling, data monitoring and statistical analyses were supervised by the Coordinating Center for Clinical Trials (KKS) of Philipps-University of Marburg; data quality and safety principles were applied. Additionally an independent Data Safety Monitoring Board was nominated. Randomisation occured and was controlled centrally through the randomisation's central office in KKS Marburg. The current study qualifies as a single-blinded trial. Assessment interviews are conducted and analyzed by people blinded to the treatment condition. Treatments in the previous randomized controlled trial were manualized, and therapists received an intense training. Treatment fidelity/integrity were analyzed with rating schemes for an priori defined proportion of randomly selected videotaped treatment sessions. Allowed additional treatments during study inclusion were thoroughly monitored and analyzed.

The sample size calculation was based on the primary outcome variable "somatization severity index" of the Screening of Somatoform Disorders (SOMS-7T). Based on results of the main validation study of SOMS-7T, metaanalytic estimations, and results of a pilot study of the efficacy of ENCERT, the power calculations yield a necessary total sample size of N=194 to detect a clinical relevant difference of 4 points symptom reduction on SOMS-7T between the two treatments with a power of 0.80 and an alpha=.05. With regard to an estimated drop-out rate of 25%, N=255 patients were recruited.

As main efficacy analysis the primary outcome shall be analyzed with linear mixed-effect models according to the ITT principle. Multilevel longitudinal mediation analyses will be conducted in order to test whether the effect of treatment condition on intraindividual changes in somatic symptom severity can be explained by intraindividual changes in emotion regulation skills.

ELIGIBILITY:
Inclusion Criteria (are based on DSM-5 diagnosis "somatic symptom disorder [SSD] 300.82"):

* Multiple distressing somatic symptoms (≥ 3 symptoms) not fully explained by a medical condition
* Pain Disability Index (mPDI) total score ≥ 4
* Patient Health Questionnaire-15 (PHQ-15) ≥ 5
* Requested psychological criteria for SSD (at least 1 of 3):

  1. Disproportionate and persistent thoughts about the seriousness of one's symptoms
  2. Persistently high level of anxiety about health or symptoms
  3. Excessive time and energy devoted to these symptoms or health concerns
* Symptom duration ≥ 6 months
* Age: 18-69 years
* Comorbidity (depression, other mental disorders) allowed, as long as somatic symptoms are considered to be the major problem by therapist and patient
* Thorough medical check for medical disease that might fully explain the somatic symptoms
* Documented medical evaluation

Exclusion Criteria:

* Severe alcohol/drug addiction
* Acquired brain injuries
* Psychoses (history of schizophrenia spectrum disorders; bipolar disorders)
* Primary disorder requesting other treatments (e.g., suicidality)
* Biomedical etiology of major symptoms (also if detected during treatment course
* Ongoing psychotherapy
* Continuous or intermittent, high-dosage (on average more than once per 2 weeks) benzodiazepine treatment
* Continuous antipsychotic treatment
* Continuous opioid treatment
* For patients on medication with antidepressants: treatment regime changes during the time between 4 weeks prior to treatment until follow-up

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in somatic symptom severity (Screening of Somatoform Disorders, SOMS-7T) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of somatic symptom severity during the last 7 days (self-rating)

SECONDARY OUTCOMES:
Change in depressive symptoms (Beck Depression Inventory-II, BDI-II) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of depressive symptoms (self-rating)
Change in emotion regulation skills (Emotion Regulation Skills Questionnaire, ERSQ) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of emotion regulation skills (self-rating)
Change in symptom-focused coping strategies (Pain Coping Questionnaire) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of symptom-focused coping strategies (self-rating)
Change in general psychopathological symptoms (Symptom Checklist-90, SCL-90) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of general psychopathological symptoms (self-rating)
Change in symptom-caused disability (Pain Disability Index, PDI) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of symptom-caused disability in different areas of life (self-rating)
Change in health-related quality of life (EuroQoL-5D, EQ-5D) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of health-related quality of life (self-rating)
Change in health anxiety (modified Short Health Anxiety Inventory, mSHAI) from pre-assessment to 3-year follow-up | From pre-assessment (admission) to follow-up (42 months after admission)
  Assessment of health anxiety (self-rating)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kleinstäuber, PhD, Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data sharing statement Will individual participant data be available (including data dictionaries)? Yes
  What data in particular will be shared? Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
  What other documents will be available? Study protocol
  With whom? Researchers who provide a methodologically sound proposal for re-analyses
  For what types of analyses? For re-analyses if their aim is covered by the purpose described and agreed on in the patient information sheet and informed consent.
Supporting Information: Study Protocol
Time Frame: Immediately following publication; no end date
Access Criteria: Proposals should be directed to the corresponding author (MK; maria.kleinstaeuber@staff.uni-marburg.de). To gain access, data requestors will need to sign a data access agreement. Data are not publicly available because informed consent provided by participants of this study is committed to a defined purpose.